CLINICAL TRIAL: NCT06119321
Title: Evaluation of a Novel Scheimpflug Device for Detection of Early Keratoconus
Brief Title: A Study of a Novel Scheimpflug Device in Diagnosing Keratoconus
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023026
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Scansys; Pentacam; Corvis ST; Keratoconus; Subclinical Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal control group
  Interventions: Other: Pentacam, Corvis ST and Scansys
- Subclinical keratoconus
  Interventions: Other: Pentacam, Corvis ST and Scansys
- Keratoconus
  Interventions: Other: Pentacam, Corvis ST and Scansys

INTERVENTIONS:
Other: Pentacam, Corvis ST and Scansys — morphological and biomechanical parameters of corneal were obtain by Scansys, Pentacam and Corvis ST

SUMMARY:
Comparison of the screening and diagnosis ability of the novel Scheimpflug-based tomography device (Scansys) with Pentacam and the Scheimpflug-based biomechanics device (Corvis ST) for keratoconus.

ELIGIBILITY:
Inclusion criteria:

* Best corrected visual acuity (BCVA) ≥ 20/20;
* No other eye diseases except myopia and astigmatism;
* The cornea was transparent, and there was no cloud or pannus;

Exclusion Criteria:

* The presence of ocular diseases other than myopia and keratoconus;
* Ocular trauma;
* Previous ocular surgery;
* Patients were required to stop wearing soft contact lenses for at least 2 weeks and rigid contact lenses for at least 4 weeks before examination;
* Pregnant and lactating women;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients premedicated for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
screening and diagnosis ability | one year
  Calculate the cut-off values, sensitivity and specificity of parameters measured by Pentacam, Corvis ST and Scansys in diagnosing keratoconus. Use Receiver operating characteristic curves (ROC) to analyze the optimal parameters to distinguish between the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided